CLINICAL TRIAL: NCT01756846
Title: Cost-effectiveness Study of the HEART Score in the Management of Patients With Chest Pain Presenting in the Emergency Room
Brief Title: Impact on Management of the HEART Risk Score in Chest Pain Patients
Acronym: HEART-Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, A.W. Hoes, Professor of Clinical Epidemiology & General Practice and Chair, Julius Center for Health Sciences and Primary Care, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 80-82310-97-12154
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Chest Pain
Keywords: HEART score; risk score; impact; chest pain
MeSH Terms: conditions — Chest Pain; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: this is a stepped wedge cluster randomized trial, meaning it is both parallel and cross-over. During 14 months, patients presenting with chest pain to the ED of participating hospitals will be included in the study. First, all hospitals will apply 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital will sequentially start to apply the HEART score in all chest pain patients (intervention period).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (Other): Daily practice of the cardiologist or attending emergency doctor, in order to diagnose a patient with chest pain. In this period attending doctors assess the risk of a patient with chest pain, based on his/hers experience and various criteria (for example described in European Society of Cardiology Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation, without a formal risk score).
  Interventions: Other: usual care
- use of HEART risk score (Other): see intervention
  Interventions: Other: use of HEART risk score

INTERVENTIONS:
Other: usual care — During 14 months, patients presenting with chest pain to the ED of participating hospitals will be included in the study. First, all hospitals will apply 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital will sequentially start to apply the HEART score in all chest pain patients (intervention period); during this intervention period patients with a HEART score 0-3 will not be admitted to the hospital, and patients with a HEART score above 3 will be treated according to current guidelines.
  Arms: usual care
Other: use of HEART risk score — During 14 months, patients presenting with chest pain to the ED of participating hospitals will be included in the study. First, all hospitals will apply 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital will sequentially start to apply the HEART score in all chest pain patients (intervention period); during this intervention period patients with a HEART score 0-3 will not be admitted to the hospital, and patients with a HEART score above 3 will be treated according to current guidelines.
  Arms: use of HEART risk score

SUMMARY:
Aim of this study is to quantify the impact of the use of the HEART risk score on patient outcome and on costs in patients with chest pain presenting at the emergency room, as compared to not using the score.

DETAILED DESCRIPTION:
During 14 months, patients presenting with chest pain to the Emergency Department (ED) of participating hospitals will be included in the study. First, all hospitals will apply 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital will sequentially start to apply the HEART score in all chest pain patients (intervention period); during this intervention period patients with a HEART score 0-3 will not be admitted to the hospital (in accordance with the results of our validation studies), and patients with a HEART score above 3 will be treated according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with chest pain to the (cardiac) ED of ten participating Dutch hospitals, older than 18 years.

Exclusion Criteria:

* Children (age <18 years) are excluded from study participation. Subjects who are (for whatever reason) not able to fill in questionnaires are excluded from study participation. Legal incapacity of every patient will be assessed by the attending doctor, according to the guidelines of legal incapacity. In case of doubt, consultation of the cardiologist (primary local investigator) will be possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3666 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arno W Hoes, MD, PhD, Principal Investigator — UMC Utrecht
Locations (9):
- Netherlands (9):
  - Amstelland Hospital, Amstelveen
  - VU Medical Center, Amsterdam
  - Gelderse Vallei, Ede
  - Catharina Hospital, Eindhoven
  - Atrium Medical Center, Heerlen
  - St. Antonius Hospital, Nieuwegein
  - Diakonessenhuis, Utrecht
  - University Medical Center, Utrecht
  - Zuwe Hofpoort, Woerden

IPD SHARING:
Plan to Share IPD: Undecided
No plans, always interested in collaboration

REFERENCES:
- [Background] Backus BE, Six AJ, Kelder JH, Gibler WB, Moll FL, Doevendans PA. Risk scores for patients with chest pain: evaluation in the emergency department. Curr Cardiol Rev. 2011 Feb;7(1):2-8. doi: 10.2174/157340311795677662. PMID 22294968
- [Background] Backus BE, Six AJ, Kelder JC, Mast TP, van den Akker F, Mast EG, Monnink SH, van Tooren RM, Doevendans PA. Chest pain in the emergency room: a multicenter validation of the HEART Score. Crit Pathw Cardiol. 2010 Sep;9(3):164-9. doi: 10.1097/HPC.0b013e3181ec36d8. PMID 20802272
- [Background] Six AJ, Backus BE, Doevendans PA. Rapid diagnostic protocol for patients with chest pain. Lancet. 2011 Jul 30;378(9789):398; author reply 398-9. doi: 10.1016/S0140-6736(11)61204-X. No abstract available. PMID 21803199
- [Background] Six AJ, Backus BE, Kingma A, Kaandorp SI. Consumption of diagnostic procedures and other cardiology care in chest pain patients after presentation at the emergency department. Neth Heart J. 2012 Dec;20(12):499-504. doi: 10.1007/s12471-012-0322-6. PMID 23090421
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Nieuwets A, Poldervaart JM, Reitsma JB, Buitendijk S, Six AJ, Backus BE, Hoes AW, Doevendans PA. Medical consumption compared for TIMI and HEART score in chest pain patients at the emergency department: a retrospective cost analysis. BMJ Open. 2016 Jun 16;6(6):e010694. doi: 10.1136/bmjopen-2015-010694. PMID 27311905
- [Background] Poldervaart JM, Reitsma JB, Koffijberg H, Backus BE, Six AJ, Doevendans PA, Hoes AW. The impact of the HEART risk score in the early assessment of patients with acute chest pain: design of a stepped wedge, cluster randomised trial. BMC Cardiovasc Disord. 2013 Sep 26;13:77. doi: 10.1186/1471-2261-13-77. PMID 24070098
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Result] Poldervaart JM, Reitsma JB, Backus BE, Koffijberg H, Veldkamp RF, Ten Haaf ME, Appelman Y, Mannaerts HFJ, van Dantzig JM, van den Heuvel M, El Farissi M, Rensing BJWM, Ernst NMSKJ, Dekker IMC, den Hartog FR, Oosterhof T, Lagerweij GR, Buijs EM, van Hessen MWJ, Landman MAJ, van Kimmenade RRJ, Cozijnsen L, Bucx JJJ, van Ofwegen-Hanekamp CEE, Cramer MJ, Six AJ, Doevendans PA, Hoes AW. Effect of Using the HEART Score in Patients With Chest Pain in the Emergency Department: A Stepped-Wedge, Cluster Randomized Trial. Ann Intern Med. 2017 May 16;166(10):689-697. doi: 10.7326/M16-1600. Epub 2017 Apr 25. PMID 28437795
- [Result] Poldervaart JM, Langedijk M, Backus BE, Dekker IMC, Six AJ, Doevendans PA, Hoes AW, Reitsma JB. Comparison of the GRACE, HEART and TIMI score to predict major adverse cardiac events in chest pain patients at the emergency department. Int J Cardiol. 2017 Jan 15;227:656-661. doi: 10.1016/j.ijcard.2016.10.080. Epub 2016 Oct 30. PMID 27810290
- See also: official website of the HEART risk score — http://www.heartscore.nl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion at 9 Dutch Emergency departments, recruitment period between 1-7-2013 and 31-8-2014.
Pre-assignment Details: Exclusion criteria were evident ST-segment elevation myocardial infarction, language barriers, recurrent presentation, or unable or unwilling to give informed consent.
Groups:
- Usual Care: usual care was defined as daily practice of the cardiologist or attending emergency doctor, in order to diagnose a patient with chest pain. In this period attending doctors assess the risk of a patient with chest pain, based on his/hers experience and various criteria (for example described in European Society of Cardiology Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation, without a formal risk score).
- HEART Care: HEART care: usual care, complemented by calculation of the HEART score and following the recommended policy.
  During 14 months, patients presenting with chest pain to the emergency department (ED) of participating hospitals were included in the study. First, all hospitals applied 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital sequentially started to apply the HEART score in all chest pain patients (intervention period); during this intervention period patients with a HEART score 0-3 were advised not be admitted to the hospital, and patients with a HEART score above 3 were advised to be treated according to current guidelines.
Period: Overall Study
Arm/Group | Usual Care | HEART Care
Started | 1833 | 1833
Completed | 1827 | 1821
Not Completed | 6 | 12
Not completed — Lost to Follow-up | 5 | 10
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: standard care of the cardiologist according to current cardiological guidelines
- HEART Care: standard care of the cardiologist according to current cardiological guidelines, complemented by calculation of the HEART score and following the recommended policy
- Total: Total of all reporting groups
Arm/Group | Usual Care | HEART Care | Total
Number analyzed (Participants) | 1827 | 1821 | 3648
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 62 (14) | 62 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 822 | 846 | 1668
  Male | 1005 | 975 | 1980
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 1827 | 1821 | 3648

OUTCOME MEASURES:

1. Primary Outcome: MACE (Major Adverse Cardiac Events)
Description: occurrence of major adverse cardiac events (MACE, i.e. acute myocardial infarction (AMI), Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Grafting (CABG) or death) within 6 weeks after presentation
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- HEART Care: HEART care: usual care, complemented by calculation of the HEART score and following the recommended policy.
Arm/Group | Usual Care | HEART Care
Number analyzed (Participants) | 1827 | 1821
Participants | 405 | 345

2. Secondary Outcome: Cost-effectiveness (Costs, QoL, QALYs)
Description: Information on quality of life (QoL) and costs was collected in 5 of the 9 hospitals. Costs for health care resource use were calculated based on Dutch guidelines and cost tables for hospitals. Different costs were used for academic and general hospitals, and costs were adjusted for inflation by using the consumer price indices provided by Statistics Netherlands. For each patient the costs were calculated based on the observed number and type of health care resources used and the type of hospital (academic/general). Data on resource use were collected for each patient in the 5 hospitals; no data were missing. QoL was derived from the EQ-5D-3L questionnaire, consisting of 5 questions (dimensions) with 3 answers each, from which QoL scores (utility values, 0-1, the higher the better) can be directly derived. Quality-adjusted life-years (scale 0-100, higher the better) were calculated over a period of 3 months, based on the estimated QoL values at 0 weeks, 2 weeks, and 3 months.
Time Frame: 3 months
Population: Cost-effectiveness analysis was performed in 5 of 9 hospitals
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Usual Care | HEART Care
Number analyzed (Participants) | 1176 | 804
years | 0.16 [0.16 to 0.17] | 0.17 [0.17 to 0.18]

3. Other Pre Specified Outcome: Gender-related Differences in Risk for MACE
Description: with a women-specific questionnaire, we hope to identify risk factors specific for women (pregnancy diabetes/hypertension, Poly Cystic Ovarial Syndrome (PCOS), etc)
Time Frame: 3 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Pre-specified Subgroup Analyses
Description: To assess whether the effectiveness and/or safety of using the HEART (history, ecg, age, risk factors, troponin) score (scale 0-10, with higher scores meaning a higher risk on MACEs) is different between specific patient populations, the following pre-specified subgroup analyses will be performed: Age: below and above 62 years of age (median), Gender: Men vs Women, Diabetics vs non-diabetics, Ethnicity: Caucasian vs. other ethnicity.
  RESULTS: None of the pre-specified subgroup analyses of women, elderly patients, and diabetic patients showed a statistically significantly different effect of HEART care with respect to incidence of MACEs. Ethnicity was unfortunately not possible to analyse due to too much missing data.
  NB. I am currently not working in the organisation which has the data, and this will not be possible the coming period. Therefore, I cannot provide correct numbers currently on these subgroup analyses, only conclusions. I am sorry for this inconvenience.
Time Frame: 6 weeks
Reporting Status: Not Posted, anticipated posting 2019-01

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- HEART Care: HEART care: usual care, complemented by calculation of the HEART score and following the recommended policy.
  During 14 months, patients presenting with chest pain to the ED of participating hospitals were included in the study. First, all hospitals applied 'usual care' to all patients, i.e. risk assessment and subsequent management without application of the HEART score. Then, during a 14 month period, each 1,5 month 1 randomly allocated hospital sequentially started to apply the HEART score in all chest pain patients (intervention period); during this intervention period patients with a HEART score 0-3 were advised not be admitted to the hospital, and patients with a HEART score above 3 were advised to be treated according to current guidelines.
Arm/Group | Usual Care | HEART Care
All-Cause Mortality (participants affected / at risk) | 9/1827 | 5/1821
Serious Adverse Events (participants affected / at risk) | 405/1827 | 345/1821
Other Adverse Events (participants affected / at risk) | 0/1827 | 0/1821
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=1827) | HEART Care (N=1821)
Cardiac ischemia (Cardiac disorders) | 400 (400) | 329 (329)
Death (Cardiac disorders) | 9 (9) | 5 (5)
Significant stenosis (PCI, CABG, conservative) (Cardiac disorders) | 290 (290) | 247 (247)

LIMITATIONS AND CAVEATS:
Hesitance to refrain from admission and testing in patients with low scores could explain the low impact on health care costs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No